CLINICAL TRIAL: NCT04110184
Title: Haematological Indices in Systemic Lupus Erythematosus and Their Association With Disease Activity
Brief Title: Haematological Indices in Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AA Mohamed, doctor, Assiut University
Other Study IDs: Haematological indices
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Rheumatic Diseases; Systemic Lupus Erythematosus
MeSH Terms: conditions — Rheumatic Diseases; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- active systemic lupus erythematosus
  Interventions: Other: Systemic lupus erythematosus disease activity index (SLEDAI)
- inactive systemic lupus erythematosus
  Interventions: Other: Systemic lupus erythematosus disease activity index (SLEDAI)

INTERVENTIONS:
Other: Systemic lupus erythematosus disease activity index (SLEDAI) — The SLEDAI score ranges between 0 and 105, and scores ≥8 represent active disease

SUMMARY:
The aim of this study is to investigate the value of several hematological indices such as:

* neutrophil-lymphocyte ratio.
* platelet-lymphocyte ratio.
* red blood cell distribution width.
* mean platelet volume (MPV), RDW/platelet ratio.
* neutrophil / C3 ratio.
* All these as biomarkers of activity in systemic lupus erythematosis patients.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a clinically common autoimmune disease characterized by abnormal immune response to autologous tissue, eventually resulting in systemic disorders and diverse clinical manifestations of the patients.

The pathogenesis of SLE remains unclear, but environmental triggers and genetic factors contribute to the destruction of immune tolerance systems, the production of immunological lymphocytes, antibodies, and inflammatory cytokines.

The clinical manifestations of SLE range from constitutional symptoms, such as fever, sweats, weight loss, joint pain and skin rashes (including the classic butter fly rash), to more serious features, including the involvement of the central nervous system and kidneys.

However, to make a clinical diagnosis of SLE, The SLICC criteria require either that a patient satisfy at least 4 of 17 criteria, including at least 1 of the 11 clinical criteria and one of the six immunologic criteria, or that the patient has biopsy-proven nephritis compatible with SLE in the presence of antinuclear antibodies (ANA) or anti-double-stranded DNA (dsDNA) antibodies. Patients with higher disease activity often present severer damage of tissues and organs.

SLE is characterized by high heterogeneity, a complex pathophysiology and various clinical manifestations; thus, no test alone is sufficiently sensitive or specific for diagnosis. Active and inactive SLE patients were evaluated according to SLE disease activity index (SLEDAI).There is significant interest in the identification of biomarkers that can predict SLE and quantify disease activity.

Neutrophils and lymphocytes play major roles in inflammatory processes. Under inflammatory conditions, neutrophil and lymphocyte counts undergo temporary changes. Neutrophil to lymphocyte ratio (NLR) is calculated as the absolute count of neutrophils divided by the absolute count of lymphocytes.

As an index of systemic inflammation, NLR has been identified to be a useful index for the differential diagnosis or prognostic prediction of diseases. NLR can be calculated easily and less costly as compared with detection of other inflammatory cytokines that could be used as biomarkers for inflammatory response or disease activity in SLE patient.

The platelet-to-lymphocyte ratio (PLR), red blood cell distribution width (RDW), and similar parameters [ eg, neutrophil-to-lymphocyte ratio (NLR) and mean platelet volume (MPV) ], which can be easily obtained using peripheral blood parameters, have been regarded as novel, accurate inflammatory biomarkers in many diseases.

MPV is a biomarker of platelet turnover, whereas platelet activation is a marker of inflammation. Previous studies have reported that MPV is correlated with the inflammatory process and disease activity in RA and ankylosing spondylitis, but the relationship between MPV and SLE remains controversial.

Complement system activation, production and partial deposition of complement fragments, and subsequent inflammation all play critical roles in the pathogenesis of SLE. During the complement activation pathway, Complement 3 was at the core position.

ELIGIBILITY:
Inclusion Criteria:

* 1. SLE patients who fulfills the 2012 Systemic Lupus International Collaborating Clinics (SLICC) criteria (Petri et al., 2012).
* 2. All patients > 18 years old.

Exclusion Criteria:

* 1. Patients with other autoimmune disease such as: Rheumatoid arthritis (RA), Mixed connective tissue disease (MTCD), Dermatomyositis (DM) and Systemic Sclerosis (SS).
* 2. Patients with malignant diseases.
* 3. Patients with coronary artery disease, cerebrovascular disease, renal and liver diseases.
* 4. Patients with evidence of any concomitant inflammatory disease. Acute infection or chronic inflammatory status.
* 5. Patients with hematological disease or history of blood transfusion in the previous 4 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 42 systemic lupus patients divided into two groups. The first group with active disease and the second group with inactive. There are 42 healthy participants age and sex matched as control group.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
hematological indices and their association with activity in systemic lupus erythematosis patients. | baseline
  investigate the value of several hematological indices and their association with activity in systemic lupus erythematosis patients.

REFERENCES:
- [Background] Gordon C, Amissah-Arthur MB, Gayed M, Brown S, Bruce IN, D'Cruz D, Empson B, Griffiths B, Jayne D, Khamashta M, Lightstone L, Norton P, Norton Y, Schreiber K, Isenberg D; British Society for Rheumatology Standards, Audit and Guidelines Working Group. The British Society for Rheumatology guideline for the management of systemic lupus erythematosus in adults: Executive Summary. Rheumatology (Oxford). 2018 Jan 1;57(1):14-18. doi: 10.1093/rheumatology/kex291. No abstract available. PMID 29029296
- [Background] Gorial FI (2018) A Clinical Utility of Neutrophil Lymphocyte Ratio as A Prognostic Indicator of Systemic Lupus Erythematosus Disease Activity. J. Pharm. Sci. & Res. 10(3) : 637-639.
- [Background] La Paglia GMC, Leone MC, Lepri G, Vagelli R, Valentini E, Alunno A, Tani C. One year in review 2017: systemic lupus erythematosus. Clin Exp Rheumatol. 2017 Jul-Aug;35(4):551-561. Epub 2017 Jul 11. PMID 28721860
- [Background] Bombardier C, Gladman DD, Urowitz MB, Caron D, Chang CH. Derivation of the SLEDAI. A disease activity index for lupus patients. The Committee on Prognosis Studies in SLE. Arthritis Rheum. 1992 Jun;35(6):630-40. doi: 10.1002/art.1780350606. PMID 1599520
- [Background] Petri M, Orbai AM, Alarcon GS, Gordon C, Merrill JT, Fortin PR, Bruce IN, Isenberg D, Wallace DJ, Nived O, Sturfelt G, Ramsey-Goldman R, Bae SC, Hanly JG, Sanchez-Guerrero J, Clarke A, Aranow C, Manzi S, Urowitz M, Gladman D, Kalunian K, Costner M, Werth VP, Zoma A, Bernatsky S, Ruiz-Irastorza G, Khamashta MA, Jacobsen S, Buyon JP, Maddison P, Dooley MA, van Vollenhoven RF, Ginzler E, Stoll T, Peschken C, Jorizzo JL, Callen JP, Lim SS, Fessler BJ, Inanc M, Kamen DL, Rahman A, Steinsson K, Franks AG Jr, Sigler L, Hameed S, Fang H, Pham N, Brey R, Weisman MH, McGwin G Jr, Magder LS. Derivation and validation of the Systemic Lupus International Collaborating Clinics classification criteria for systemic lupus erythematosus. Arthritis Rheum. 2012 Aug;64(8):2677-86. doi: 10.1002/art.34473. PMID 22553077
- [Background] Yu H, Jiang L, Yao L, Gan C, Han X, Liu R, Su N. Predictive value of the neutrophil-to-lymphocyte ratio and hemoglobin insystemic lupus erythematosus. Exp Ther Med. 2018 Aug;16(2):1547-1553. doi: 10.3892/etm.2018.6309. Epub 2018 Jun 13. PMID 30112073
- [Background] Yu J, Zeng T, Wu Y, Tian Y, Tan L, Duan X, Wu Q, Li H, Yu L. Neutrophil-to-C3 ratio and neutrophil-to-lymphocyte ratio were associated with disease activity in patients with systemic lupus erythematosus. J Clin Lab Anal. 2019 Jan;33(1):e22633. doi: 10.1002/jcla.22633. Epub 2018 Aug 20. PMID 30129188
- [Background] Xie S, Chen X. Red blood cell distribution width-to-platelet ratio as a disease activity-associated factor in systemic lupus erythematosus. Medicine (Baltimore). 2018 Sep;97(39):e12342. doi: 10.1097/MD.0000000000012342. PMID 30278511
- [Background] Qin B, Ma N, Tang Q, Wei T, Yang M, Fu H, Hu Z, Liang Y, Yang Z, Zhong R. Neutrophil to lymphocyte ratio (NLR) and platelet to lymphocyte ratio (PLR) were useful markers in assessment of inflammatory response and disease activity in SLE patients. Mod Rheumatol. 2016;26(3):372-6. doi: 10.3109/14397595.2015.1091136. Epub 2016 Mar 4. PMID 26403379
- [Background] Balta S, Aparci M, Ozturk C, Demirkol S, Celik T. Neutrophil-lymphocyte ratio as an useful mortality marker. Am J Emerg Med. 2014 Dec;32(12):1546-7. doi: 10.1016/j.ajem.2014.09.040. Epub 2014 Oct 2. No abstract available. PMID 25315881
- [Background] Safak S, Uslu AU, Serdal K, Turker T, Soner S, Lutfi A. Association between mean platelet volume levels and inflammation in SLE patients presented with arthritis. Afr Health Sci. 2014 Dec;14(4):919-24. doi: 10.4314/ahs.v14i4.21. PMID 25834502
- [Result] Ayna AB, Ermurat S, Coskun BN, Harman H, Pehlivan Y. Neutrophil to Lymphocyte Ratio and Mean Platelet Volume as Inflammatory Indicators in Systemic Lupus Erythematosus Nephritis. Arch Rheumatol. 2016 Aug 17;32(1):21-25. doi: 10.5606/ArchRheumatol.2017.5886. eCollection 2017 Mar. PMID 30375538